CLINICAL TRIAL: NCT03364816
Title: Evaluation on Efficacy of Total Artificial Disc Replacement (TDR) of Cervical Spondylosis: a Cohort Prospective Follow-up for 5 Years
Brief Title: Evaluation on Efficacy of Total Artificial Disc Replacement (TDR) of Cervical Spondylosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Zhenqi, Clinical Professor, Peking University People's Hospital
Other Study IDs: TDR
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Cervical Spondylosis
Keywords: cervical spondylosis; artificial disc replacement; complications; photographic indicators; functional efficacy
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TDR with Prodisc-C: participant underwent total disc replacement with Prodisc-C artificial disc
  Interventions: Procedure: TDR
- TDR with Mobi-C: participant underwent total disc replacement with Mobi-C artificial disc
  Interventions: Procedure: TDR
- TDR with Prestige-LP: participant underwent total disc replacement with Prestige-LP artificial disc
  Interventions: Procedure: TDR

INTERVENTIONS:
Procedure: TDR — total artificial disc replacement

SUMMARY:
To evaluate the efficacy of 3 different types of cervical disc prosthesis (Prodisc-C, Mobi-C and Prestige-LP) in the treatment of cervical spondylosis.

DETAILED DESCRIPTION:
A cohort, retrospective analysis will be performed of 150 patients who were in implementation of artificial disc replacement in our department from 2008 to 2012 and accepted a regular postoperatively follow-up up to 5 years, the sample will be divided into 3 groups according to prosthesis and 50 people in each group. The outcome will be measured among 3 groups respectively on the operation (such as operation time, intraoperative bleeding.), postoperative complications (such as prosthesis sinking, displacement and prolapse, adjacent segments degeneration and heterotopic ossification), photographic indicators and functional efficacy analysis and then a comparison for self-contrast pre- and post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients was diagnosed as cervical spondylosis based on imaging and symptomology;
2. patients were purely underwent TDR within the three kinds of prosthesis;
3. the range of participants is from 20-65 years;
4. conservative treatment of 6 months is invalid;
5. never had cervical operations.

Exclusion Criteria:

1. Patients suffered from cervical trauma or congenital malformations;
2. non-artificial cervical disc replacement or hybrid surgery;
3. ones who refused to be followed up.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. The range of participants is from 20-65 years;
  2. conservative treatment of 6 months is invalid;
  3. never had cervical operations;
  4. operation on one to three segments.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
JOA score | 5 years
  The whole name is Japanese Orthopaedic Association Scores for Assessment of Cervical spondylosis, the range of JOA is 0-17 and the full score is 17 to represent a normal function.

SECONDARY OUTCOMES:
prosthesis sinking | 5 years
  prosthesis sinking is defined by a sink of 2mm about the artificial disk postoperatively.
range of motion (ROM) | 5 years
  range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Zhu, Principal Investigator — Department of spinal surgery

IPD SHARING:
Plan to Share IPD: No